CLINICAL TRIAL: NCT00823953
Title: The Effect of Momordica Charantia on Glycemic Control and Insulin Resistance in Type 2 Diabetes
Brief Title: Glycemic Response to Momordica Charantia in Type 2 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IP could not be made available in sufficient quantity for the expected enrollment
Sponsor: Services Hospital, Lahore (Other Government)
Collaborators: University of the Punjab (Other)
Responsible Party: Principal Investigator, Khadija Irfan Khawaja, Assistant Professor of Endocrinology, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMC0107
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: diabetes type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo powder (wheat flour) The placebo arm will be administered capsules containing a total of 500 mg of starch powder, at dose level 1; 1000 mg at dose level 2; 1500 mg at dose level 3.
  Interventions: Other: starch powder
- Momordica charantia (Active Comparator): Thirty patients will be assigned to each arm in a double blind manner. The active arm will be administered capsules containing a total of 500 mg of Momordica charantia freeze dried powder, at dose level 1; 1000 mg at dose level 2; 1500 mg at dose level 3.
  The placebo arm will be administered capsules containing a total of 500 mg of starch powder, at dose level 1; 1000 mg at dose level 2; 1500 mg at dose level 3.
  Interventions: Drug: Momordica charantia

INTERVENTIONS:
Drug: Momordica charantia — escalating doses of Momordica charantia administered in the form of capsules for the trial phase of three week.Dose level 1: capsules containing a total of 500 mg of freeze dried powder of Momordica charantia. Dose level 1: capsules containing a total of 1000 mg of freeze dried powder of Momordica charantia. Dose level 3: capsules containing a total of 1500mg of freeze dried powder of Momordica charantia.
  Other Names: Bitter Melon Capsule
  Arms: Momordica charantia
Other: starch powder — The placebo arm will be administered capsules containing a total of 500 mg of starch powder, at dose level 1; 1000 mg at dose level 2; 1500 mg at dose level 3.
  Arms: Placebo

SUMMARY:
Diabetes is a common disease which has been treated by traditional medicines for centuries before modern medicine became available. A very common remedy for Diabetes Mellitus in different cultures is momordica charantia (karela or Bitter gourd). The use of alternative medicine is common among Pakistani population. This study was planned to find out the effect of administering freeze dried powder of momordica charantia for three weeks on the glycemic profile and insulin resistance of treatment naiive patients with mild Type 2 diabetes.

DETAILED DESCRIPTION:
Momordica charantia is a commonly consumed vegetable, which has formed a part of subcontinental diet since centuries. It has been traditionally used to treat diabetes across three continents, and its glycemic effect has been investigated in a few unblinded trials, but so far no properly designed double blind investigation of its action on insulin resistance has not been carried out. In this study, a randomised placebo controlled double-blind trial will be carried out on mild type 2 diabetic patients, to study the effect of escalating doses of Momordica charantia administered in the form of capsules for the trial phase of three weeks, on glycemic control and parameters of insulin resistance in type 2 diabetes. Among the parameters to be tested will be glucose indices and lipid profile and insulin levels. The effect of Momordica charantia administration on insulin resistance will be assessed using HOMA-IR model and/ or the hyperinsulinemic, euglycemic clamp. The selection of patients with mild hyperglycemia will be done to offset the glucose spill-off effect which occurs beyond the real threshold, and makes the glucose tolerance curve non-linear beyond this level.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Type 2 diabetics with mild degree of hyperglycemia (FBG >126<200 mg/dl)
2. Absence of serious co-morbid conditions
3. Patients agreeing to participate in this trial

Exclusion Criteria:

1. Type 1 diabetics
2. Pregnancy
3. Paediatric age group
4. Patients known to be allergic to Momordica charantia
5. Serious cardio-respiratory illness, previous myocardial infarction, angina pectoris, heart failure, uncontrolled hypertension ≥ stage 2, COPD, asthma, active pulmonary tuberculosis
6. Significant hepatic impairment: ALT >60, Bilirubin >2 mg/dl
7. Significant renal impairment: S/creatinine >1.5 mg/dl, albuminuria > 1+
8. Patients with conditions likely to interfere with the absorption of the trial therapy: malabsorption, chronic diarrhoea, intestinal resection, blind loop syndrome
9. Patients withholding consent
10. Patients, both male and female, desiring pregnancy during the trial phase.
11. Secondary causes of diabetes
12. Patients using drugs influencing glucose metabolism: steroids, hormonal contraception, menopausal HRT , diazoxide, phenytoin, colchicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
serum fructosamine at end of trial phase in each of the groups | three weeks

SECONDARY OUTCOMES:
Development of major adverse effects (e.g. intractable vomiting, jaundice, allergic reactions or other effects requiring cessation of therapy and breaking of study code) | three weeks
GLP-1[7-36] in each group at the end of trial phase | three weeks
FBG at end of trial phase in each of the groups | three weeks
HOMA-IR in each of the two groups at end of trial phase | three weeks
Insulin resistance by the hyperinsulinemic, euglycemic clamp in a subset at the end of trial phase | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khadija I Khawaja, MBBS,FCPS, Principal Investigator — Services Hospital, Lahore
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Ahmed I, Adeghate E, Sharma AK, Pallot DJ, Singh J. Effects of Momordica charantia fruit juice on islet morphology in the pancreas of the streptozotocin-diabetic rat. Diabetes Res Clin Pract. 1998 Jun;40(3):145-51. doi: 10.1016/s0168-8227(98)00022-9. PMID 9716917
- [Background] Ahmed I, Lakhani MS, Gillett M, John A, Raza H. Hypotriglyceridemic and hypocholesterolemic effects of anti-diabetic Momordica charantia (karela) fruit extract in streptozotocin-induced diabetic rats. Diabetes Res Clin Pract. 2001 Mar;51(3):155-61. doi: 10.1016/s0168-8227(00)00224-2. PMID 11269887
- [Background] Dans AM, Villarruz MV, Jimeno CA, Javelosa MA, Chua J, Bautista R, Velez GG. The effect of Momordica charantia capsule preparation on glycemic control in type 2 diabetes mellitus needs further studies. J Clin Epidemiol. 2007 Jun;60(6):554-9. doi: 10.1016/j.jclinepi.2006.07.009. Epub 2006 Nov 13. PMID 17493509
- See also: Database File for Momordica charantia — http://www.rain-tree.com/bitmelon.htm